CLINICAL TRIAL: NCT05884463
Title: 18F-FAPI PET/CT and 18F-FDG PET/CT in Patients With Pancreatic Adenocarcinoma : A Prospective, Single-Center, Comparative Study
Brief Title: 18F-FAPI PET Imaging in Pancreatic Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPIPDAC01
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: 18F-FAPI; 18F-FDG; Pancreas Adenocarcinoma; Diagnosis; Staging
MeSH Terms: conditions — Disease | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients underwent both 18F-FDG PET/CT and 18F-FDG PET/CT scan
  Interventions: Drug: 18F-FAPI; Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FAPI — Intravenous injection of one dosage of 18F-FAPI.
  Other Names: (18)F-FAPI
Drug: 18F-FDG — Intravenous injection of one dosage of 18F-FDG.
  Other Names: (18)F-FDG

SUMMARY:
To explore the potential efficacy of 18F-FAPI-04 PET/CT for PDAC tumour staging and compare the results with those obtained using 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Accurate diagnosis and staging are crucial for selecting treatment for patients with pancreatic ductal adenocarcinoma (PDAC). The desmoplastic responses associated with PDAC are often characterised by hypometabolism. Here we investigated 18F-fibroblast activation protein inhibitor (18F-FAPI-04) positron emission tomography/computed tomography (PET/CT) in evaluation of PDAC, and compared the findings with those obtained using (18F)-fluorodeoxyglucose (18F-FDG).

ELIGIBILITY:
Inclusion Criteria:

patients who were suspected to have PDAC by radiological imaging patients who underwent paired 18F-FAPI-04 PET/CT and 18F-FDG PET/CT for metastasis screening, recurrence confirmation, or tumour staging patients who were willing to participate in clinical trials and signed an informed consent form.

Exclusion Criteria:

patients with a history of severe contrast allergy pregnant patients patients who were not pathologically diagnosed as showing PDAC.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic value | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  Sensitivity and Specificity of 18F-FAPI PET/CT for diagnosis and staging in comparison with 18F-FDG PET/CT
Maximum standardized uptake value | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  SUVmax of 18F-FAPI PET/CT for lesions in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Diagnostic efficacy for primary lesions | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  Sensitivity, specificity, accuracy of 18F-FAPI PET/CT for primary lesions in comparison with 18F-FDG PET/CT
SUVmax for primary lesions | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  SUVmax of 18F-FAPI PET/CT for primary lesions in comparison with 18F-FDG PET/CT
SUVmax for lymph node | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  SUVmax of 18F-FAPI PET/CT for lymph node in comparison with 18F-FDG PET/CT
SUVmax for distant metastasis | 1 day (At the time the patient has underwent both 18F-FAPI and 18F-FDG PET/CT)
  SUVmax of 18F-FAPI PET/CT for distant metastasis in comparison with 18F-FDG PET/CT
Correlation between the SUVmax of 18F-FAPI and 18F-FDG uptake in patients with different treatment response | at least 2 months after treatment
  The correlation of SUVmax and treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Ph.D., M.D., Study Director — Zhejiang University
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Li X, Lu N, Lin L, Chen Y, Yang S, Wang H, Liu X, Wu C, Xue X, Su X, Bai X, Liang T. 18F-FAPI-04 Outperforms 18F-FDG PET/CT in Clinical Assessments of Patients with Pancreatic Adenocarcinoma. J Nucl Med. 2024 Feb 1;65(2):206-212. doi: 10.2967/jnumed.123.266283. PMID 38176719